CLINICAL TRIAL: NCT05810350
Title: The Efficacy and Safety of Aumolertinib Combined Ommaya Reservoir Intrathecal Chemotherapy With Pemetrexed for Leptomeningeal Metastasis From EGFR-mutated NSCLC and Investigate the Efficacy Prognostic Value of Dynamic Changes of cfDNA
Brief Title: Aumolertinib Combined Intrathecal Chemotherapy for Leptomeningeal Metastasis From EGFR-Mutated NSCLC and Prognostic Value of Dynamic Changes in cfDNA Profiles
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Three Gorges Hospital of Chongqing University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022(No.166)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR; cfDNA; leptomeningeal metastasis; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: Aumolertinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aumolertinib combined Ommaya reservoir intrathecal chemotherapy (Experimental): Aumonertinib 165mg orally once daily and intrathecal chemotherapy with pemetrexed (30 mg was administered on days 1 and 8) once every 3 weeks.
  Interventions: Drug: Aumonertinib 165mg orally once daily and intrathecal chemotherapy with pemetrexed

INTERVENTIONS:
Drug: Aumonertinib 165mg orally once daily and intrathecal chemotherapy with pemetrexed — Patients receive Aumonertinib 165mg orally once daily and intrathecal chemotherapy with pemetrexed (30 mg was administered on days 1 and 8) once every 3 weeks.

SUMMARY:
This is a prospective, open-label, single-arm clinical trial. The aim of this study is to evaluate the efficacy and safety of almonertinib and intrathecal chemotherapy in patients with advanced EGFR mutation positive (EGFRm+) non-small cell lung cancer (NSCLC) and leptomeningeal metastasis, and to explore the predictive value of dynamic changes of cfDNA in cerebrospinal fluid for efficacy and prognosis. A total of 40 subjects who met the inclusion criteria were enrolled in the study and received almonertinib (165mg, oral, once a day) combined with intrathecal infusion. Before and after treatment, cerebrospinal fluid was extracted for cfDNA detection by a 49 gene detection panel. Treatment continued until disease progression or other discontinuation criteria were met. In addition, the subjects received regular hematological and imaging examinations to evaluate the condition. Finally, through data analysis, the progression-free survival (PFS), disease control rate (DCR), objective response rate (ORR), duration of response (DoR), and overall survival (OS) of patients with EGFR mutation-positive advanced NSCLC and leptomeningeal metastasis who received almonertinib combined with intrathecal infusion chemotherapy were evaluated. The dynamic changes of cfDNA in cerebrospinal fluid before and after treatment were explored and the correlation between the dynamic changes of cfDNA in cerebrospinal fluid and the therapeutic effect was explored.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single-arm clinical trial to explore the efficacy and safety of almonertinib and intrathecal chemotherapy in patients with advanced NSCLC and leptomeningeal metastasis and the predictive value of cfDNA changes for efficacy and prognosis. A total of 40 patients aged 18 years or older with confirmed advanced NSCLC with leptomeningeal metastases and an EGFR sensitive mutation (exon 19 deletion or 21 L858R) are expected to be enrolled. The intervention was almonertinib (165mg orally, once daily) combined with intrathecal infusion therapy (pemetrexed 30 mg by injection on days 1 and 8 of each cycle). Treatment continued until disease progression or other discontinuation criteria were met.

Relevant examinations and data collection during the study were as follows. CSF collection: Approximately 15mL of CSF was collected from each sample, and sampling was performed before C1D1 administration and within one week after PD (24 hours after the previous day's administration). Venous blood sample collection: subjects who underwent CSF sampling were performed before C1D1 and C2D1 administration (24 hours after the previous day's dose) and within 1 week after PD. Before treatment, all enrolled patients underwent neurological examination, complete blood count, serum biochemistry, coagulation indexes, blood tumor markers, cytological and CSF tumor markers, electrocardiogram, brain and spinal cord MRI, chest and abdominal CT, and bone scan. The blood and CSF tests described above were performed for each treatment cycle. Imaging was performed every 2 months or if clinical progression was suspected until death. Before each intrathecal infusion, LM-related neurological symptoms, PS score, Neuro-oncology Working Group (RANO) score, and headache score were assessed and recorded in detail. Adverse events (AEs) were graded and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).

The primary objective was to evaluate the progression-free survival (PFS) of almonertinib versus intrathecal chemotherapy in patients with advanced EGFR mutation-positive NSCLC and leptomeningeal metastases. The secondary study objectives were: first, to evaluate the efficacy of almonertinib and intrathecal chemotherapy in the treatment of advanced NSCLC with leptomeningeal metastases: disease control rate (DCR), objective response rate (ORR), duration of response (DoR), and overall survival (OS); Intracranial: intracranial progression-free survival (iPFS), intracranial disease control rate (iDCR), intracranial objective response rate (iORR), and intracranial duration of response (iDoR). Second, evaluate the time to symptom improvement of almonertinib versus intrathecal chemotherapy in patients with EGFR mutation-positive advanced NSCLC and leptomeningeal metastases. Third, we evaluated the safety of almonertinib and intrathecal infusion chemotherapy in patients with EGFR mutation-positive advanced NSCLC and leptomeningeal metastases. The objectives of this pilot study were as follows: 1) To evaluate the correlation between baseline and post-treatment cfDNA changes in CSF and treatment response; Second, the correlation between baseline CSF cfDNA status and patient prognosis; Third, sensitivity analysis based on baseline CSF cfDNA mutations and leptomeningeal metastases after targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old.
* The Eastern Cancer Organization Collaboration Group (ECOG) had a physical fitness score of 0 to 3, and had not worsened in the previous 2 weeks, with a minimum expected survival of 12 weeks.
* NSCLC confirmed by histology or cytology, positive cerebrospinal fluid cytology, and combined with central nervous system function and brain imaging findings, diagnosed as NSCLC with meningeal metastasis (including advanced patients who had relapsed or were initially diagnosed after previous surgical treatment; GPA is recommended for grading and typing in the diagnosis of meningeal metastasis from lung cancer).
* Tumor tissue samples or blood samples were tested and confirmed as EGFR sensitive mutations (including exon 19 deletion or L858R, both alone or coexisting with other EGFR site mutations). The first choice is to submit tumor tissue for examination; If the tumor tissue is inaccessible or the subject is not eligible for tissue biopsy, a blood sample may be sent for examination.
* The patient has implanted an Ommaya capsule;
* CT examination of clinical symptom areas (spine and/or brain) and/or head within the past 3 months to rule out contraindications to cerebrospinal fluid examination;
* The subjects agreed to provide two cerebrospinal fluid samples (before treatment and within one week after disease progression) for genetic testing;
* Women of childbearing age need to take appropriate contraceptive measures and should not breastfeed three months after screening and discontinuing study treatment. "Before starting administration, the pregnancy test was negative, or one of the following criteria was met to demonstrate that there was no risk of pregnancy:

  1. Postmenopause is defined as amenorrhea at least 12 months after age greater than 50 years and cessation of all exogenous hormone replacement therapy.
  2. Women younger than 50 years of age may also be considered postmenopausal if they have amenorrhea for 12 months or more after stopping all exogenous hormone therapy, and their luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels are within the laboratory postmenopausal reference values.
  3. Have undergone irreversible sterilization surgery, including hysterectomy, bilateral ovariectomy, or bilateral salpingectomy, except for bilateral tubal ligation.
* Male subjects should use barrier contraception (i.e., condoms) three months after screening and discontinuation of study treatment.
* The subject voluntarily participated and signed an informed consent form in writing.

Exclusion Criteria:

* Have received any of the following treatments:

  1. Within 4 weeks before the first administration of the investigational drug, the subject had undergone major surgery (such as craniotomy, thoracotomy, or laparotomy). The definition of major surgical surgery refers to Level 3 and Level 4 surgery specified in the "Management Measures for Clinical Application of Medical Technology" implemented on November 1, 2018;
  2. Within 7 days before the first administration of the study drug, a strong CYP3A4 inhibitor, inducer, or CYP substrate (CYP2C8, CYP2D6, etc.) was used.
  3. Subjects with other malignant tumors, excluding basal cell carcinoma of the skin and carcinoma in situ.
* At the beginning of the study treatment, there was a residual toxicity greater than CTCAE level 3 that could not be alleviated from previous treatment.
* There are pleural effusion/peritoneal effusion requiring clinical intervention (patients who do not require drainage of the effusion or who have been stable for 2 weeks or more after drainage can be enrolled); Presence of pericardial effusion (small amounts of pericardial effusion that are stable for 2 weeks or more are allowed to be included in the group). If local use (such as thoracic perfusion) of anti-tumor drugs is used during drainage, and at least 5 drug half-lives or 21 days (whichever is shorter) must be eluted before the first administration of the study treatment before enrollment;
* Subjects are unwilling to provide cerebrospinal fluid samples or clinical information;
* Subjects have contraindications for cerebrospinal fluid examination;
* Previously or currently suffering from primary malignant tumors of the central nervous system;
* Suffering from autoimmune or inflammatory diseases of the central nervous system (not limited to multiple sclerosis, neurosarcoidosis, chronic fungal, rickettsial, or bacterial meningitis);
* Subjects who are allergic to the MRI contrast agent gadolinium or who cannot tolerate MRI examination (such as having a cardiac pacemaker, having metal in their body, etc.).
* According to the judgment of the researcher, there are any serious or poorly controlled systemic diseases, such as poorly controlled hypertension, active hemorrhagic constitution, or active infection. There is no need to screen for chronic diseases.
* Clinically severe gastrointestinal dysfunction may affect the intake, transportation, or absorption of drugs, such as inability to take orally, uncontrollable nausea or vomiting, a history of extensive gastrointestinal resection, untreated recurrent diarrhea, atrophic gastritis, untreated stomach diseases requiring long-term administration of mass pump inhibitors, Crohn's disease, ulcerative colitis, and so on.
* Hepatic encephalopathy, hepatorenal syndrome, or cirrhosis.
* Meet any of the following cardiac examination results:

  1. The mean value of the QT interval (QTcF) corrected by Fridericia's formula from three electrocardiogram (ECG) examinations at rest is>470 msec;
  2. resting ECG indicates conduction or ECG morphological abnormalities (such as complete left bundle branch block, 3rd degree atrioventricular block, 2nd degree atrioventricular block, and PR interval>250 msec);
  3. The presence of any factors that increase the risk of QTc prolongation or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome, or any concomitant medication that causes unexplained sudden death or prolongs the QT interval in immediate family members under the age of 40;
  4. Left ventricular ejection fraction (LVEF)<50%.
* Insufficient bone marrow reserve or organ function, reaching any of the following laboratory limits (no corrective treatment within 1 week before laboratory examination and blood sampling):

  1. Absolute neutrophil count<1.5 × 109 / L；
  2. Platelet count<100 × 109 / L；
  3. Hemoglobin<90 g/L (<9 g/dL);
  4. If there is no clear liver metastasis, alanine aminotransferase is>3 times the upper normal limit (ULN); If there is liver metastasis, alanine aminotransferase>5 × ULN；
  5. If there is no clear liver metastasis, aspartate aminotransferase>3 × ULN； If there is liver metastasis, aspartate aminotransferase>5 × ULN；
  6. If there is no clear liver metastasis, total bilirubin>1.5 × ULN； Or presence of Gilbert syndrome (unconjugated hyperbilirubinemia) or liver metastasis with total bilirubin>3 × ULN；
  7. Creatinine>1.5 × ULN and creatinine clearance<50 mL/min (calculated using the Cockcroft Gault formula); Only when creatinine>1.5 × It is only necessary to confirm the creatinine clearance rate at ULN;
  8. Serum albumin (ALB)<28 g/L.
* Active fungal, bacterial, and/or viral infections that require systemic treatment.
* Female subjects who are pregnant, nursing, or planning to become pregnant during the study period.
* Have a history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of radiation pneumonia requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
* A history of hypersensitivity to any active or inactive component of aumolertinib, or to drugs with a chemical structure similar to or in the same category as aumolertinib.
* Patients who are allergic to or contraindicated to pemetrexed.
* Any serious or uncontrolled ocular lesions (especially severe dry eye syndrome, dry corneal conjunctivitis, severe exposure keratitis, or other diseases that may increase epithelial damage) that, in the judgment of a doctor, may increase the safety risk of the subject; Or eye abnormalities that require surgery or are expected to require surgical treatment during the study period.
* Subjects who, according to the judgment of the investigator, may have poor compliance with the research procedures and requirements, such as having a clear history of neurological or mental disorders (including epilepsy or dementia), or currently suffering from mental disorders.
* The investigator determines that there are any conditions that endanger the safety of the subject or interfere with the evaluation of the study, or other conditions that the researcher believes are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 18 months.
  PFS is defined as the time from date of enrollment until the date of disease progression as assessed according to RECIST 1.1 or death from any cause on study.

SECONDARY OUTCOMES:
intracranial progress free survival | 18 months.
  iPFS is defined as the time from date of enrollment until the date of disease progression in intrathecal lesions as assessed according to Response Assessment in Neuro-Oncology or death from any cause on study.
objective response rate | 18 months.
  ORR is defined as the number of patients with at least 1 visit response of CR (Complete response) or PR (Partial response) according to RECIST 1.1.
Disease control rate | 18 months.
  Disease control rate (DCR) is defined as the percentage of participants with disease control best overall response (complete response, partial response or stable disease).
overall survival | From baseline until death due to any cause,up to a maximum of approximately 3 years.
  OS is defined as time from date of enrollment until date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
Incidence of Adverse Events (AEs) | From the screening period to 28 days after treatment completion, approximately 3 years.
  AEs are graded according to CTCAE v5.0 and recorded in the case report form.

CONTACTS AND LOCATIONS:
Locations (1):
- chongqing University Three Gorges Hospital, Chongqing, China